CLINICAL TRIAL: NCT04796207
Title: Study of Effect of Docosahexaenoic Acid (DHA) and Eicosapentaenoic Acid (EPA) Supplementation on Biomarkers of Sub-Concussion Injuries in American Football
Brief Title: The Effects of Fish Oil Supplementation on the Brain Health of Collegiate Football Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Floyd Chilton, Professor, Department of Nutritional Sciences Director, Precision Nutrition & Wellness Initiative Associate Director,The BIO5 Institute, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB1904553365
Record Dates: First submitted 2021-03-03; First posted 2021-03-12 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Traumatic Brain Injury (TBI); Chronic Traumatic Encephalopathy (CTE)
Keywords: CTE (Chronic Traumatic Encephalopathy); mTBI (Mild Traumatic Brain Injury); Concussion; MRI; Nf-L (Neurofilament Light Chain); Biomarker; Football
MeSH Terms: conditions — Brain Injuries, Traumatic; Chronic Traumatic Encephalopathy; Brain Concussion; Charcot-Marie-Tooth disease, Type 1F | interventions — Fish Oils; Capsules

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to treatment (3 grams DHA and EPA (2:1 weight ratio)) or placebo (3 grams high-oleic safflower oil in a 1:1 allocation ratio) based on their position on the football team and roster depth (starter vs. non-starter). Participants will be recruited as a single cohort. After screening, participants will be treated with DHA and EPA or matching placebo for 25 weeks (a full course of an American football season, including summer camp training sessions). A follow-up visit is scheduled 7 weeks after the final dosing at week 32 for recovery and adverse event evaluation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study personnel will be kept blind to treatment assignments. The treatment assignment for each participant will be available to the investigator in a sealed envelope that may be opened only in the case of a serious adverse event which the investigator feels cannot be adequately treated without knowing the identity of the study medication. Code breakers will be collected and reviewed at the end of the study. If the blinding has been broken, then the investigator will provide documentation regarding the fact and indicate the other staff that received this information.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fish Oil Capsules (Experimental): Participants in the treatment arm will receive 3 grams of DHA and EPA (2:1 weight ratio) 5 times a week for 25-weeks during regular football season.
  Interventions: Dietary Supplement: Fish Oil (DPA+EPA 2:1 ratio) Capsules
- Safflower Oil Capsules (Placebo Comparator): Participants in the treatment arm will receive 3 grams of high-oleic safflower oil (in a 1:1 allocation ratio) 5 times a week for 25-weeks during regular football season.
  Interventions: Dietary Supplement: High Oleic Safflower Oil Capsules

INTERVENTIONS:
Dietary Supplement: Fish Oil (DPA+EPA 2:1 ratio) Capsules — The Treatment Arm intervention consists of providing participants with 3 grams of DHA and EPA (2:1 weight ratio) in capsular form. In order to meet the required 3 grams of DHA and EPA, participants were given 6 capsules to be taken with meals (preferably breakfast, although capsules were provided at lunch when they couldn't be provided at breakfast). Capsules were given 5 times a week during the regular football season.
  Arms: Fish Oil Capsules
Dietary Supplement: High Oleic Safflower Oil Capsules — The Placebo Arm intervention consists of providing participants with 3 grams of high-oleic safflower oil in a 1:1 allocation ratio in capsular form. In order to maintain the "study masking", participants in the Placebo Arm were given 6 capsules (the same as the Treatment Arm) to be taken with meals (preferably breakfast, although capsules were provided at lunch when they couldn't be provided at breakfast). Capsules were given 5 times a week during the regular football season.
  Arms: Safflower Oil Capsules

SUMMARY:
Determine if the daily docosahexaenoic acid (DHA)/eicosapentaenoic acid (EPA) supplement will reduce serum levels of biomarkers of sub-concussion injuries over a course of American football season among collegiate football athletes.

DETAILED DESCRIPTION:
American football is one of the most popular sports in the U.S. Yet this sport is associated with increased risk of concussion (also known as mild traumatic brain injury, or mTBI) and sub-concussive injury from repeated head impacts (RHI) due to the aggressive and high-speed nature of the game. Current protective equipment used by players are not sufficient to reduce concussion incidence and severity, nor are there any therapeutics available to prevent concussion. This study is a randomized, double-blind, placebo controlled trial to determine if an omega-3 polyunsaturated fatty acid (PUFA) fish oil supplement containing 3.0 grams of docosahexaenoic acid (DHA; 22:6n-3) and eicosapentaenoic acid (EPA; 20:5n-3) can reduce blood biomarkers of sub-concussion injuries compared to placebo (high-oleic safflower oil) over a course of the American football season among collegiate football athletes.

The dosage of DHA/EPA used in this study is generally safe, and procedures involved, monthly blood draws, surveys, and Magnetic Resonance Imaging (MRI), pose minimal risks to participants. While this study provides no direct benefit to participants, successful outcomes of this study can benefit the society by shedding light on development of potential preventative therapeutics for sports-induced mTBI and brain injury from RHI. The risk-benefit profile is appropriate for conducting this study. Based on preclinical studies and previous clinical study results, the investigators expect that in comparison to placebo treatment, DHA and EPA treatment throughout the course of one American football season can maintain lower levels of sub-concussion associated biomarkers, inflammatory cytokines, and cardiovascular risk markers. The investigators also expect participants treated with DHA and EPA to have lower brain MRI imaging markers of sub concussion injury.

ELIGIBILITY:
Inclusion Criteria:

1) University of Arizona National Collegiate Athletic Association (NCAA) Division I American football athletes cleared to participate in university athletics as determined by the team physician.

Exclusion Criteria:

1. Chronic daily anti-inflammatory drugs (>20 d).
2. Medications for blood lipids.
3. Active fish oil or omega-3 fatty acid supplementation.
4. Consumption of more than two servings of fish per week.
5. Injured and unable to participate in regularly schedule conditioning or competitions.
6. Acute concussion experienced within 30 days of starting the study.
7. Fish allergies.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Age: 18-25 Gender: Male Ethnicity: All races and ethnicities
Enrollment: 38 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Floyd Chilton, Ph.D., Principal Investigator — University of Arizona; Roberta Brinton, Ph.D., Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

REFERENCES:
- [Derived] Raikes AC, Hernandez GD, Mullins VA, Wang Y, Lopez C, Killgore WDS, Chilton FH, Brinton RD. Effects of docosahexaenoic acid and eicosapentaoic acid supplementation on white matter integrity after repetitive sub-concussive head impacts during American football: Exploratory neuroimaging findings from a pilot RCT. Front Neurol. 2022 Sep 15;13:891531. doi: 10.3389/fneur.2022.891531. eCollection 2022. PMID 36188406

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fish Oil Capsules | Safflower Oil Capsules
Started | 19 | 19
Completed | 12 | 17
Not Completed | 7 | 2
Not completed — Lost to Follow-up | 7 | 2

BASELINE CHARACTERISTICS:
Population: NCAA football participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Fish Oil Capsules | Safflower Oil Capsules | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 38
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.9 (0.70) | 21.2 (2.07) | 21.05 (1.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 19 | 19 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 14 | 25
  Not Hispanic or Latino | 8 | 5 | 13
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Changes in Brain Biomarkers Due to Sub-concussion Injury - Nf-L
Description: This primary outcome covers the change in the plasma brain biomarker Neurofilament Light Chains (Nf-L) due to sub-concussion injury from baseline to predetermined measurement time points. Nf-L (neuron specific intermediate proteins) are released upon injury to neurons and axons. Measured in picograms per milliliter (pg/ml)
Time Frame: Baseline, Week 17, Week 26
Measure: Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Fish Oil Capsules | Safflower Oil Capsules
Number analyzed (Participants) | 12 | 17
pg/ml
  Baseline | 5.36 [4.71 to 6.00] | 4.82 [4.54 to 5.10]
  Week 17 | 6.05 [5.65 to 6.44] | 6.47 [6.14 to 6.8]
  Week 26 | 7.61 [6.54 to 8.69] | 6.21 [5.86 to 6.57]

2. Primary Outcome: Changes in Sub-concussion Injury Related Inflammation Biomarkers - TNF-α
Description: This primary outcome covers the change in the plasma inflammation biomarker Tumor Necrosis Factor-alpha (TNF-α), a cytokine and mediator of inflammation, due to sub-concussion injury from baseline to predetermined measurement time points. TNF-α is measured in picograms per milliliter (pg/ml).
Time Frame: Baseline ans Week 26
Measure: Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Fish Oil Capsules | Safflower Oil Capsules
Number analyzed (Participants) | 12 | 17
pg/ml
  Baseline | 1.181 [1.02 to 1.34] | 0.962 [0.91 to 1.01]
  Week 26 | 1.039 [0.86 to 1.22] | 0.918 [0.88 to 0.96]

3. Primary Outcome: Changes in Sub-concussion Injury Related Inflammation Biomarkers - IL-6
Description: This primary outcome covers the change in the plasma inflammation biomarker Interleukin-6 (IL-6), a cytokine and mediator of inflammation, due to sub-concussion injury from baseline to predetermined measurement time points. IL-6 is measured in picograms per milliliter (pg/ml)
Time Frame: Baseline; Week 17; Week 26
Measure: Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Fish Oil Capsules | Safflower Oil Capsules
Number analyzed (Participants) | 12 | 17
pg/ml
  Baseline | 2.186 [1.71 to 2.66] | 1.309 [1.12 to 1.50]
  Week 17 | 2.338 [1.77 to 2.90] | 2.107 [1.71 to 2.50]
  Week 26 | 2.158 [1.52 to 2.79] | 1.761 [1.53 to 1.99]

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events were reported to study staff daily when supplements were delivered.
Arm/Group | Fish Oil Capsules | Safflower Oil Capsules
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/17
Other Adverse Events (participants affected / at risk) | 12/12 | 11/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fish Oil Capsules (N=12) | Safflower Oil Capsules (N=17)
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 9 (9) — Common cold
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
GI distress (Gastrointestinal disorders) | 3 (3) | 0 (0) — Stomach upset
Halitosis (Gastrointestinal disorders) | 4 (4) | 0 (0) — Bad breath
Concussion (Nervous system disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT04796207/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/07/NCT04796207/SAP_001.pdf